CLINICAL TRIAL: NCT00731848
Title: An Open-label Extension Study of the Effects of Pomegranate Extract on Rising Prostate-specific Antigen Levels in Men Following Primary Therapy for Prostate Cancer.
Brief Title: Open-label Extension Study of the Effects of Pomegranate Extract on Rising PSA After Primary Therapy for Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Roll International Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUP-0205-1X
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate-specific antigens; PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Intervention 1
  Interventions: Dietary Supplement: pomegranate liquid extract

INTERVENTIONS:
Dietary Supplement: pomegranate liquid extract — Pomegranate liquid extract, 8 oz per day, for 52 weeks

SUMMARY:
This study is an open-label extension to the double-blind GUP-0205-1 and double-blind extension GUP-0205-1XX studies. High concentrations of anti-oxidants in pomegranate seeds present a potential strategy to delay clinical prostate cancer progression and prolong the interval from treatment failure to hormonal ablation. Eligible male subjects were previously assigned to the placebo group in the double-blind core study or the double-blind extension study and were diagnosed with disease progression while on placebo treatment. Upon satisfying all entry criteria, the subjects will receive open-label pomegranate extract for up to 48 months in the absence of further disease progression or intolerable toxicity.

DETAILED DESCRIPTION:
This study is an open-label extension to the double-blind GUP-0205-1 and double-blind extension GUP-0205-1XX studies. Eligible male subjects, i.e.,men who had rising PSA levels following primary therapy for localized prostate cancer, were previously assigned to the placebo group in the double-blind study or the double-blind extension and were diagnosed with disease progression while on placebo treatment. Upon satisfying all entry criteria, the subjects will receive open-label pomegranate extract for up to 48 months in the absence of further disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Documented disease progression while on placebo in the GUP-0205-1 or GUP-0205-1XX study (a ≥100% increase over baseline serum PSA with a minimum increase of 1.0 ng/mL.
* Willingness and ability to sign an informed consent document.
* Agreement with complete abstinence from other commercially available pomegranate products during the course of the study.
* Use of dietary/herbal supplements (e.g., saw palmetto, selenium, etc) are acceptable provided the dose has been stable for at least 2 months prior to screening and the subject agrees not to change/stop during the course of the study.
* Performance status 0 or 1 on the ECOG scale at time of entry into this extension Study.

Exclusion Criteria:

* Significant concomitant medical or psychiatric condition that, in the opinion of the investigator, would make the subject a poor protocol candidate.
* Hormonal therapy, with the exception of neoadjuvant androgen deprivation therapy (ADT) prior to or concurrent with primary therapy. Subjects who underwent neoadjuvant ADT cannot have a serum testosterone of ≤150 ng/mL at study entry.
* Concomitant or antecedent hormonal therapy for rising serum PSA after initial therapy of prostate cancer.
* Subjects unable or unwilling to comply with protocol requirements.
* Prior treatment with experimental drugs, high dose steroids, or with any other cancer treatment within 4 weeks prior to the first dose of study product and for the duration of the study.
* Serum PSA >7.0 ng/mL (assessed at termination of the double-blind study or ET of the double-blind extension GUP-0205-1XX); at any PSA level, the subject will be excluded if determined by the investigator that the subject's continued participation would not be in their best interest).
* Serum PSA doubling time <13 weeks (assessed at termination of the double-blind study or ET of the double-blind extension GUP-0205-1XX)).
* Evidence of metastatic disease on physical examination or on CT or bone scan.
* Use of finasteride, dutasteride at any point since primary therapy or during the study.
* Clinically significant abnormal laboratory value greater than 2 times the upper limit of normal (>2XULN).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
The within-subject difference between the PSA doubling time from the end of double-blind placebo treatment to the end of open-label pomegranate extract treatment. | 12 months

SECONDARY OUTCOMES:
The effect of treatments on response rates for positive PSA doubling times (greater than 150% baseline), and for negative post-treatment PSA doubling time (i.e., declining PSA), and for changes in absolute PSA values. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan J Pantuck, MD, Principal Investigator — University of California, Los Angeles; Arie S Belldegrun, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA School of Medicine, Los Angeles, California, United States